CLINICAL TRIAL: NCT03279900
Title: Hematotoxicity in Acute Lymphoblastic Leukemia Children in Maintenance Phase Therapy at Cipto Mangunkusumo Hospital and Its Affecting Factors
Brief Title: Hematotoxicity in Acute Lymphoblastic Leukemia Children in Maintenance Phase Therapy
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dewi Selvina Rosdiana, Researcher at Department of Pharmacology and Therapeutics Faculty of Medicine University of Indonesia, Indonesia University
Other Study IDs: IndonesiaUI
Record Dates: First submitted 2017-08-28; First posted 2017-09-12 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study use an observational study design from patient medical records to obtain data on patient demographics, nutritional status, 6MP dosing, and albumin levels of LLA child patients.

DETAILED DESCRIPTION:
All medical record data of LLA child patient at maintenance phase therapy, who came to Cipto Mangunkusumo Kiara Hospital in period 2014 - 2016. the data that are colected consist of age, gender, disease stratification, nutritional status, the dosage of 6-MP, albumin levels, hemoglobin levels, leukocyite counts, platelet counts, and absolute neutrophil counts.

ELIGIBILITY:
Medical record of Acute Limphoblastic Leukemia patients at Cipto Mangunkusumo Hospital, in period of 2012 - 2014, with Inclusion Criteria:

* LLA Patients, male and female, age 1 - <18 years
* Received chemotherapy maintenance phase based on Indonesian protocol of ALL - 2013

Exclusion Criteria:

* Incomplete medical record data.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Medical record of Acute Limphoblastic Leukemia patients at Cipto Mangunkusumo Hospital, in period of 2012 - 2014
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
The Incidence of hematotoxicity in acute limphoblastic leukemia children during maintenance phase therapy. | october 2017
  based on medical record data: Incidence of anemia, Neutropenia, and thrombocytopenia in acute limphoblastic leukemia children during maintenance phase therapy.

SECONDARY OUTCOMES:
The relationship of the incidence of hematotoxicity with influencing factors | November 2017
  The relationship of the incidence of hematotoxicity (anemia, Neutropenia, thrombocitopenia) with ALL stratification (High risk or Standard risk, as written in the medical record), nutritional status (normal or malnutrition), and albumin levels (normal or Hypoalbuminemia). The determination of nutritional status is based on body weight (Kg) and Height (Meters). Determination of nutritional status using cutoff Z score based on The growth chart of WHO 2006 for children 0-5 years, and ideal weight percentage according to Waterlow criteria for children above 5 years (recommendation of Indonesian Pediatric Association).

CONTACTS AND LOCATIONS:
Overall Officials: Rianto Setiabudy, Professor, Study Director — Departemen of Pharmacology and therapeutics, FMUI
Locations (1):
- Cipto Mangunkusomo hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No